CLINICAL TRIAL: NCT07407790
Title: The Southern-Norway Post-Stroke Atrial Fibrillation Study
Acronym: SNAPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: REKID 931942
Record Dates: First submitted 2026-01-25; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF); Atrial Fibrillation (Prevention of Stroke); Ischemic Stroke; Secondary Prevention; Arrhythmia Atrial
Keywords: stroke; atrial fibrillation; anticoagulation
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, parallel-group, open-label (no masking) screening study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (ECG247 Smart Heart Sensor) (Experimental): Patients in this group will have the ECG247 patch applied to the anterior chest wall while in the hospital.
  * Device: The ECG247 is a wireless, water-resistant patch sensor that connects to a dedicated smartphone application via Bluetooth. It transmits data to a secure cloud service for analysis.
  * Duration: The device is worn continuously for up to 14 days. Monitoring begins in-hospital and continues after discharge.
  * Analysis: The system utilizes an algorithm to detect arrhythmia. Episodes of AF >30 seconds are considered positive findings. Study personnel and physicians verify algorithm-detected episodes.
  * Concurrent Care: These patients also receive standard in-house telemetry per hospital protocol while admitted.
  Interventions: Device: Patch ECG
- Control Arm (Standard Care) (Other): Patients in this group receive standard heart rhythm monitoring according to current hospital guidelines.
  * In-hospital: Monitoring via continuous telemetry or intermittent ECGs based on availability and clinical priority.
  * Ambulatory: Upon discharge, patients are referred for ambulatory Holter monitoring. The duration is typically 24-48 hours as decided by the treating cardiologist.
  * Analysis: Holter recordings are analyzed by trained technicians and reviewed by a cardiologist.
  Interventions: Device: Standard Care (in control arm)

INTERVENTIONS:
Device: Patch ECG — This study aims to evaluate the clinical utility and cost-effectiveness of a novel, continuous patch ECG system (ECG247) initiated in the hospital setting compared to standard care.
  Arms: Intervention Arm (ECG247 Smart Heart Sensor)
Device: Standard Care (in control arm) — Patients in this group receive standard heart rhythm monitoring according to current hospital guidelines.
  Arms: Control Arm (Standard Care)

SUMMARY:
This study evaluates whether a procedure using a new wireless heart sensor patch is equal to or better than the standard hospital procedures and equipment at detecting an irregular heartbeat called Atrial Fibrillation (AF) after an ischemic stroke. Atrial fibrillation is a major cause of stroke, but it can be difficult to catch because it often comes and goes.

The study will include approximately 450 adults who have had a stroke or a transient "mini-stroke" (TIA) within the last two weeks. Participants will be assigned by chance (randomized) to one of two groups:

* Group 1 (Intervention): Participants wear the "ECG247 Smart Heart Sensor." This is a small patch that sticks to the chest and connects to a smartphone. It is worn continuously for up to 14 days, even after leaving the hospital.
* Group 2 (Standard Care): Participants receive the standard hospital check-up. This typically involves using a "Holter monitor" (a device with wires and electrodes) for a period of about 24 to 48 hours some time after leaving the hospital.

The main goal is to see if the procedure using the patch is equal to the standard procedure in detecting atrial fibrillation in participants. The study will also measure how quickly doctors can start the correct medication and how easy the patients find the devices to use.

DETAILED DESCRIPTION:
Background and Rationale Atrial fibrillation (AF) is a major risk factor for ischemic stroke, yet it often goes undetected due to its paroxysmal (intermittent) nature. While guidelines recommend prolonged heart rhythm screening after a stroke of undetermined cause, standard hospital practice often relies on short-term telemetry and ambulatory Holter monitoring. These standard methods can be limited by device availability, bulkiness, and short monitoring duration (typically 24-48 hours), potentially leading to under-diagnosis of AF.

This study aims to evaluate the clinical utility and cost-effectiveness of a novel, continuous patch ECG system (ECG247) initiated in the hospital setting compared to standard care.

Study Design This is a prospective, randomized, parallel-group, open-label (no masking) study conducted at a single stroke center. Approximately 450 eligible patients will be enrolled.

Recruitment and Stratification Patients admitted with ischemic stroke or transient ischemic attack (TIA) within the last two weeks are screened for eligibility, aiming for inclusion within 48 hours of admission. Participants are randomized in a 1:1 ratio to either the intervention arm or the standard care arm. Randomization is stratified by age into three groups: 18-64 years, 65-74 years, and ≥75 years.

Intervention Arm (ECG247 Smart Heart Sensor) Patients in this group will have the ECG247 patch applied to the anterior chest wall while in the hospital.

* Device: The ECG247 is a wireless, water-resistant patch sensor that connects to a dedicated smartphone application via Bluetooth. It transmits data to a secure cloud service for analysis.
* Duration: The device is worn continuously for up to 14 days. Monitoring begins in-hospital and continues after discharge.
* Analysis: The system utilizes an algorithm to detect arrhythmia. Episodes of AF >30 seconds are considered positive findings. Study personnel and physicians verify algorithm-detected episodes.
* Concurrent Care: These patients also receive standard in-house telemetry per hospital protocol while admitted.

Control Arm (Standard Care) Patients in this group receive standard heart rhythm monitoring according to current hospital guidelines.

* In-hospital: Monitoring via continuous telemetry or intermittent ECGs based on availability and clinical priority.
* Ambulatory: Upon discharge, patients are referred for ambulatory Holter monitoring. The duration is typically 24-48 hours as decided by the treating cardiologist.
* Analysis: Holter recordings are analyzed by trained technicians and reviewed by a cardiologist.

Biomarker Analysis Blood samples will be collected from all participants to analyze N-terminal pro-B-type natriuretic peptide (NT-proBNP) levels. The study will assess the association between NT-proBNP levels and the detection of silent AF to evaluate its potential for risk stratification.

Outcomes and Follow-up

* Primary Outcome: The detection rate of AF (defined as episodes ≥30 seconds).
* Secondary Outcomes: Time to AF detection, time to initiation of anticoagulation therapy, total monitoring duration, and health economics.
* User Experience: Patients in the intervention group will complete Patient Reported Experience Measures (PREMs) regarding usability and satisfaction.
* Long-term Follow-up: Participants will be followed for up to 12 months to assess clinical endpoints, including secondary stroke, TIA, and major bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with an ischemic stroke or transient ischemic attack (TIA), including amaurosis fugax, occurring within the last 2 weeks.
* Initial evaluation of CT and/or CT angiography and/or MRI supports a diagnosis of TIA or ischemic stroke.
* Available smartphone and access to the ECG247-app to be able to participate in the study.
* Estimated life span of >6 month
* Permanent address in Norway
* Informed Consent, Capable of giving signed informed consent or consent through proxy as described in Appendix which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the study protocol.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

* Known AF or atrial flutter prior to inclusion
* Concomitant use of anticoagulation therapy or established contraindication to its use. To date this includes apixaban, rivaroxaban, edoxaban, dabigatran, warfarin and indirect thrombin inhibitors (except for short term thrombosis prevention).
* Implanted pacemaker, ICD or loop-recorder
* >70% stenosis of carotid artery on ipsilateral side to the stroke on CT angiography or ultrasound
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate of atrial fibrillation | From enrollment to the end of heart rate monitoring. Will also be registered on follow up after 12 months.
  The detection rate of AF (defined as episodes ≥30 seconds). Analysis will be performed on an intention-to-treat basis, and AF detection will be primarily assessed for its non-inferiority and secondarily for difference in proportions. An interim analysis for efficacy measures will be performed using the O'Brien-Flemming correction for the primary endpoint AF detection rate after 72 and 144 participants in each arm.
Time from enrollment to treatment initiation with anticoagulant medicine | From enrollment until end of follow up (12 months after enrollment).
  Days from enrollment until AF detection results in change of prophylactic treatment, defined as prescribed anticoagulant medication collected by the patient, retrieved from e-prescription data accessed through the Summary Care Record (Kjernejournal).
Time from enrollment to detection of first AF episode | From enrollment up to 1 year
  Time to detection of first episode of atrial fibrillation after hospital admission
Total duration of heart rate monitoring | From enrollment up to 1 year
  Total duration of heart rate monitoring, also including an assessment of device signal quality for assessment
Numbers of participants with secondary stroke/TIA and/or major bleeding | From enrollment to one-year follow up, assessed at 1-year follow up.
  Assessing secondary stroke and major bleeding at 1 year of follow-up

SECONDARY OUTCOMES:
Explore the practical utility in regards to validity of results of AF screening after a stroke with a patch ECG | After 1 year of recruitment
  Inter-rater validity of ECG results between the ECG247 algorithm, cardiologists and neurologists
Explore the practical utility of time consumed using AF screening after a stroke with a patch ECG | After 1 year of recruitment
  A suitable number of observations will be performed to evaluate the time needed to complete the patch ECG attachment and inform the patient, interpret the results and follow-up of results
Explore the practical utility and reliability of AF screening after a stroke with a patch ECG | Assessed at 1 year after enrollment start
  Reliability of the monitoring device in crude versus interpretable monitoring duration in hours. Reliability will be assessed by the study personnel when creating the patch ECG result record. The whole pulse rate strip will be analyzed to identify periods of 1>h with a lack of signal or reduced signal quality. The total monitoring duration registered by the algorithm in hours versus manual interpretation with readable signal in hours will be evaluated as a percentage: Useable monitoring time/Total monitoring time x 100% = Percentage of useful monitoring.
Explore the practical utility and patient satisfaction of AF screening after a stroke with a patch ECG | Through study completion
  Patient Reported Experience Measures (PREMs) to all patients in interventional arm within a month of discharge and within 1 month of Holter completion for control arm, registration of technical problems, allergic reactions to patch, photo of patch placement and registration of patients not considered eligible to the study due to lack of smartphone and other causes not listed in the exclusion/inclusion criteria. PREMS will be reported by a 7 point Likert scale, with higher values indicating a high level of satisfaction.
Diagnostic quality of in-house patch ECG compared to telemetry | From start of enrollment until discharge of last included patient
  Sensitivity and specificity of AF detection in patch ECG compared to concomitant telemetry.
  Assessment of detection of other dangerous arrhythmias in patch ECG compared to telemetry.
  Quality of signal from telemetry compared to patch ECG. In the subgroup of patients where patch ECG and telemetry are worn simultaneously, the results of both methods will be cross-validated against each other
Cost effectiveness of patch ECG compared to standard care | From enrollment until end of follow up.
  Cost-effectiveness analysis of patch ECG and standard care with the endpoint being reduced secondary stroke
Assess predictors of silent AF | From enrollment until end of patient follow-up
  Association between clinical, radiological and laboratory factors (including) NT-pro-BNP level and AF NT-proBNP will be assessed upon inclusion and can be analyzed from blood samples drawn on day 1 after admission.
  MRI results Echocardiography results CHADSVASC, age, gender, medication used, previous diseases, BMI

CONTACTS AND LOCATIONS:
Locations (1):
- Sørlandet Sykehus HF, Kristiansand, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Currently undecided regarding the sharing of IPD. No established formal cooperation agreements with external research groups to date. Any future decision to share data will depend on the establishment of such collaboration agreements in adherence to data protection regulations.